CLINICAL TRIAL: NCT05327413
Title: A Prospective Cohort Study to Compare the Accuracy of Femoral External Rotation Measured on CT and MRI
Brief Title: Femoral External Rotation Measured on CT and MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, xiangshuai, Principal Investigator, The Affiliated Hospital of Qingdao University
Other Study IDs: QYFYKYLL 915211920
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Other: CT and MRI

INTERVENTIONS:
Other: CT and MRI — CT and MRI were conducted to measure the femoral external rotation

SUMMARY:
This study aims to compare the femoral external rotation measured on CT and MRI to that measured intraoperatively to clarify the influence of residual cartilage on posterior condyle on the preoperative planning of total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

1. 50-85 years old
2. patients with osteoarthritis (Kellgren-Lawrence Grade III or IV) underwent total knee arthroplasty.

Exclusion Criteria:

1. patients cannot endure TKA due to severe heart failure, arrhythmia, myocardial infarction, infection or other reason.
2. patients who cannot undergo MRI.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients underwent TKA due to knee arthroplasty (Kellgren-Lawrence Grade III or IV)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Femoral external rotation on CT | Preoperative
  the angel between the posterior condylar axis (PCA) and transepicondylar axis (TEA) on CT
Femoral external rotation on MRI | Preoperative
  the angel between the posterior condylar axis (PCA) and transepicondylar axis (TEA) on MRI
Intraoperative femoral external rotation | Intraoperative
  the angel between the posterior condylar axis (PCA) and transepicondylar axis (TEA) measured intraoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Shuai Xiang, Principal Investigator — The Affiliated Hospital of Qingdao University
Locations (1):
- The affiliated hospital of Qingdao University, Qingdao, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided